CLINICAL TRIAL: NCT05016908
Title: Extracellular RNA Biomarkers of Duchenne Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Thurman Wheeler, M.D, Physician Scientist, Massachusetts General Hospital
Other Study IDs: 2019P001504
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biofluid collection: Eligible volunteers will be asked to provide a single urine sample and undergo a single blood draw.

SUMMARY:
Current methods of measuring the response to new treatments for muscular dystrophies involve the examination of small pieces of muscle tissue called biopsies. The investigators are interested in finding less invasive methods that reduce the need for muscle biopsies. The purpose of this research is to learn about the possibility of detecting and measuring the activity and severity of muscular dystrophies by examining a urine sample and a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with DMD or BMD based on genetic testing. Control subjects are unknown to have any other muscular dystrophy by history and may have had no genetic testing.
* Able to provide informed consent or assent for participation in the study.
* Demographic characteristics for biofluid collection: Males age 5 years and older with DMD or BMD; males and females ages 18 years and older without muscular dystrophy.

Exclusion Criteria:

* Medical history of any of the following: State of immunosuppression; coagulopathy; pre-existing liver or kidney disease; documented HIV positive; documented hepatitis B and/or C positive.
* Use of anti-platelet drugs within 7 days prior to blood draw; use of anticoagulants within 60 days prior to blood draw.
* Inability or unwillingness of the subject to give written informed consent.

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Males ages 5 years and older with Duchenne muscular dystrophy (DMD) or Becker muscular dystrophy (BMD). In addition, male and female family members without known muscular dystrophy ages 18 and older also are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Extracellular RNA in biofluids | 4 years
  The extracellular RNA biomarkers in the muscular dystrophy groups will be evaluated and compared with the extracellular RNA content in control groups. Statistical analysis will be used to evaluate the sensitivity and specificity of these markers as measurements of disease activity and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Thurman M. Wheeler, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoury L, Hu N, Balaj L, Das S, Georghiou S, Darras B, Clark T, Breakefield XO, Wheeler TM. Analysis of extracellular mRNA in human urine reveals splice variant biomarkers of muscular dystrophies. Nat Commun. 2018 Sep 25;9(1):3906. doi: 10.1038/s41467-018-06206-0. PMID 30254196
- [Background] Antoury L, Hu N, Darras B, Wheeler TM. Urine mRNA to identify a novel pseudoexon causing dystrophinopathy. Ann Clin Transl Neurol. 2019 May 17;6(6):1106-1112. doi: 10.1002/acn3.777. eCollection 2019 Jun. PMID 31211175